CLINICAL TRIAL: NCT07392177
Title: An Alpha2-adrenoceptor Agonist to Reduce Locus Coeruleus Activity During Sleep in Adults With Insomnia Disorder: a Pilot Randomised Placebo-controlled Cross-over Study
Brief Title: Understanding the Role of the Locus Coeruleus in Insomnia
Acronym: LOCUSleep
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Woolcock Institute of Medical Research (Other)
Responsible Party: Principal Investigator, Christopher Gordon, Research Leader, Woolcock Institute of Medical Research
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: 19522
Record Dates: First submitted 2025-12-08; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Insomnia
Keywords: Electroencephalography; Sleep; Locus coeruleus; Hyperarousal
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Dexmedetomidine

STUDY DESIGN:
Intervention Model Description: Double-blind, randomised, placebo-controlled crossover study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All trial staff (except one unblinded researcher) and participants will be blinded to the intervention and control medication. We will use identical containers and labels except a patient identification code. The order of treatments will be secured in a password-protected data management system and known by the unblinded researcher.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dexmedetomidine (Experimental): A 96 µg dexmedetomidine tablet taken during the sleep laboratory visit only
  Interventions: Drug: Dexmedetomidine
- Placebo (Active Comparator): Matching placebo tablet taken during the sleep laboratory visit only
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dexmedetomidine — A buccal tablet containing 96 µg dexmedetomidine will be taken before habitual bedtime.
  Arms: Dexmedetomidine
Drug: Placebo — Placebo tablets will contain identical excipient without the active ingredient (dexmedetomidine) and manufactured under the same condition as the active. Placebo tablets, packs and instructions will be identical in every respect to enable the double-blind study design.
  Arms: Placebo

SUMMARY:
This research project aims to better understand the neurobiological mechanistic underpinnings of insomnia disorder. The main question is whether cortical hyperarousal in individuals with insomnia disorder, measured by electroencephalograhic (EEG) infraslow oscillation coupling of sigma power during non-rapid eye movement (NREM) sleep and theta power during rapid eye movement (REM) sleep, is related to locus coeruleus activity.

DETAILED DESCRIPTION:
This trial is a double-blinded, placebo-controlled, randomised controlled cross over trial of dexmedetomidine or placebo in adults with insomnia disorder. Participants will be recruited using social media, bulletin boards and patient referrals from the Woolcock Institute of Medical Research clinics. Participants will be asked to complete an online pre-screening webpage (RedCap) to check for eligibility, and provided with the Participant Information Sheet (PIS) and asked for contact details for an in-person screening visit. The participants will have the study explained in detail during the screening visit followed by written informed consent. The participant will then undergo a medical screening for diagnosis of insomnia disorder and the medical officer will sign the consent form. Thereafter, the participant will complete baseline questionnaires and be randomised to either dexmedetomidine or placebo for the 2 sleep laboratory visits. Participants will then be instructed to maintain their regular sleep-wake patterns for seven days before the first sleep laboratory visit (Visit 1). During Visit 1, participants will undergo a number of assessments (pre-sleep locus coeruleus activity measured using pupillometry, electroencephalography (EEG), functional near-infrared spectroscopy (fNIRS) before and during sleep and questionnaires about subjective hyperarousal. Participants will receive either dexmedetomidine or placebo. Following Visit 1, participants will have a 14-day washout, before Visit 2, which will repeat the procedures of Visit 1, but participants will receive the alternate condition (placebo or dexmedetomidine). The study will be coordinated from the Woolcock Institute of Medical Research, Sydney, Macquarie University, NSW, 2113, Australia.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of insomnia disorder (DSM-5-TR)
* Insomnia severity index (ISI) score ≥15
* Able to provide informed consent
* Fluent English literacy

Exclusion Criteria:

* Medically diagnosis of sleep disordered breathing (i.e. sleep apnea) or sleep or circadian disorder other than insomnia
* Uncontrolled psychiatric disorders
* High dependence on medical care
* History of, or current suicide ideation (Patient Health Questionnaire (PHQ-9) questionnaire)
* Pregnancy or actively trying to conceive, or lactating
* Shiftwork - defined as work outside of business hours (before 8am or after 6pm) conducted at least once per week
* Travel across time zones of over 2 h time difference in the past week
* Contraindicate the patient's participation in the clinical trial due to safety concerns or compliance with clinical study procedures
* Concomitant use of medicines that are inhibitors, or moderate to strong inducers, of CYP3A4; regular use of hypnotics and other medications that can cause additive sedation or psychostimulants or non-amphetamine psychostimulants within 14 days of starting the clinical trial
* Ongoing use of THC- or CBD-containing products; dependence or any other drug or alcohol dependence
* Allergy to lactose

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Electrographic (EEG) signatures | Baseline and 14 days
  Electrographic (EEG) infraslow oscillations (~50 sec) of sigma power and sleep spindle coupling during non-rapid eye movement (NREM) sleep and theta power during rapid eye movement (REM) sleep.

SECONDARY OUTCOMES:
Sleep Fragmentation | Baseline and 14 days
  Polysomnography (PSG) measure conducted during the intervention and control (wake after sleep onset)
EEG power | Baseline and 14 days
  Electroencephalographic (EEG) power during non-rapid eye movement (NREM) (stages 2 and 3) and rapid eye movement (REM) sleep. Unit of measurement is μV^2.
Neurovascular activity (fNIRS) | Baseline and 14 days
  Measurement of global blood flow using functional near-infrared spectroscopy (fNIRS).
Cardiopulmonary Coupling (CPC) | Baseline and 14 days
  Cardiopulmonary coupling provides a global measure of autonomic function
Pupillometry | Baseline and 14 days
  Pupil sizes will be assessed as a surrogate of locus coeruleus activity
Subjective hyperarousal | Baseline and 14 days
  Pre-Sleep Arousal Scale (PSAS) before sleep. Scored by summing 16 items (rated 1 (not at all) to 5 (extremely)) with a total score between 16 to 80
Subjective sleep quality | Baseline and 14 days
  Self-reported rating of sleep quality (0-9) with higher scores indicating worse sleep. This will assessed in the morning after the overnight sleep study.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Gordon, PhD, Principal Investigator — Woolcock Institute of Medical Research; Brendon Yee, MBChB, PhD, Principal Investigator — Woolcock Institute of Medical Research
Locations (1):
- Woolcock Institute of Medical Research, Macquarie Park, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: Yes
Non-identifiable IPD will be shared upon reasonable request to the Principal Investigators.
Supporting Information: Study Protocol, ICF, Analytic Code
Time Frame: Non-identifiable IPD will become available one year after the Actual Study Completion Date and will be available for ten years.
Access Criteria: A copy of the non-identifiable dataset may be requested by academic collaborators not affiliated with the Woolcock Institute of Medical Research through a data request form which outlines the investigators, aims and hypotheses, data to be included, a statistical analysis plan, ethics approval, and security measures. Contact the Coordinating Principal Investigator for access to data.